CLINICAL TRIAL: NCT05748171
Title: A PROSPECTIVE, RANDOMIZED, OPEN-LABEL PHASE 2 STUDY TO EVALUATE THE SUPERIORITY OF INOTUZUMAB OZOGAMICIN MONOTHERAPY VERSUS ALLR3 FOR INDUCTION TREATMENT OF CHILDHOOD HIGH RISK FIRST RELAPSE B-CELL PRECURSOR ACUTE LYMPHOBLASTIC LEUKAEMIA
Brief Title: A Study to Learn More About the Study Medicine Called Inotuzumab Ozogamicin (InO) in Children (1 to <18 Years) With First Relapse ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1931036; 2023-509810-13-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-01-20; First posted 2023-02-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: ACUTE LYMPHOBLASTIC LEUKEMIA
Keywords: ALL; BCP ALL; High risk BCP ALL; Relapse ALL; Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at 2:1 ratio, so that approximately 67 participants will receive InO and 33 participants will receive the comparator treatment regimen, ALLR3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inotuzumab ozogamicin (Experimental): Each participant in the InO arm will receive 1 course (3 doses) of InO, as follows:
  * Day 1: 0.8 mg/m2
  * Days 8 (±1 day) and Day 15 (±1 day): 0.5 mg/m2/dose
  Interventions: Drug: Inotuzumab ozogamicin
- ALLR3 (Active Comparator): Mitoxantrone 10 mg/m2 on Days 1 and 2 Vincristine 1.5 mg/m2 (max single dose 2 mg) administered on Days 3, 10, 17 and 24 Dexamethasone 20 mg/m2/day administered orally (or IV) divided into two daily doses (maximum 40 mg/day) as two 5-day blocks on Days 1-5 and Days 15-19.
  PEG-asparaginase 1000 units/m2 IV administered on Days 3 and 17. In case of hypersensitivity/allergic reaction to PEG-asparaginase, each dose of PEG-asparaginase will be replaced by Erwinia-asparaginase at a dose of 20,000 units/m² IV or IM every other day for a total of 6 doses
  Interventions: Drug: ALLR3

INTERVENTIONS:
Drug: Inotuzumab ozogamicin — Inotuzumab ozogamicin (BESPONSA™) is a CD22 targeted antibody drug conjugate (ADC) approved in several countries for the treatment of adults with relapsed or refractory B cell precursor acute lymphoblastic leukemia (ALL). The approved starting dose is 1.8mg/m2/cycle.
  Other Names: Besponsa
  Arms: Inotuzumab ozogamicin
Drug: ALLR3 — The ALLR3 chemotherapy regimen (vincristine, mitoxantrone, dexamethasone, and PEG-asparaginase [or erwinia-asparaginase in the event of an allergic reaction to PEG-asparaginase]) has been adopted by pediatric oncology groups as treatment for pediatric relapsed/refractory (R/R) acute lymphoblastic leukemia (ALL)
  Other Names: R3
  Arms: ALLR3

SUMMARY:
This prospective, randomized, multicenter, open-label Phase 2 study is designed to evaluate the superiority of InO monotherapy vs ALLR3 after 1 cycle of induction treatment in paediatric participants (between 1 and <18 years) with High Risk (HR) first bone marrow relapse CD22-positive BCP ALL, and to evaluate the safety and tolerability, PK and long-term efficacy. Treatment with study intervention will end after induction therapy; follow-up will continue for up to 5 years from randomization.

DETAILED DESCRIPTION:
This prospective, randomized, multicenter, open-label, Phase 2 study is designed to evaluate the superiority of InO monotherapy vs ALLR3, after 1 cycle of induction treatment in paediatric participants (between 1 and <18 years) with HR first bone marrow relapse CD22-positive BCP ALL, and to evaluate the safety and tolerability, PK and long-term efficacy. Treatment with study intervention will end after induction therapy; follow-up for efficacy and safety will continue for up to 5 years from randomization.

End of Treatment is defined as occurring upon recovery from 1 cycle of study therapy (Day 28 ± 2 days), or one day before initiation of new anticancer therapy, whichever occurs first.

Approximately 100 participants will be randomized (2:1) to receive 1 cycle of either InO monotherapy or ALLR3 (block 1) therapy during induction.

After completion of induction therapy (ie, study therapy), it is anticipated that the majority of responding participants will proceed immediately to consolidation therapy. Non-responders are expected to proceed with salvage therapy at the investigator's discretion. Participants responding to induction therapy are expected to proceed to SOC consolidation therapy upon recovery of blood counts, but no sooner than 7 days after last dose of study intervention.

All participants (responders and non-responders) will proceed to long-term follow-up for this study. All subsequent anticancer therapy will be determined by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between 1 and <18 years of age.
2. Morphologically confirmed diagnosis of first relapse HR BCP ALL; HR first relapse is defined as relapse occurring within 18 to 30 months of original diagnosis of ALL or within 6 months of completion of primary therapy, and lacking any identified very high-risk genetic abnormalities (Groeneveld-Krentz et al, 2019) (ie, KMT2A::AFF1 fusion [t(4;11)(q21;q23)], TCF3-HLF fusion [t(17;19)(q22;p13)], TCF3-PBX1 fusion [t(1;19)(q23;p13.3)], hypodiploidy [<40 chromosomes] or masked low hypodiploidy (Molina et al, 2021), TP53 alteration).

   * CD22-positive ALL as defined by local institution;
   * Bone marrow involvement of ≥ 5% leukemic blasts (≥ M2 status).
3. Adequate serum chemistry parameters:

   * An eGFR in participants 1 to <2 years of age, or eCrCl in those 2 to <18 years of age, ≥30 mL/min using the recommended formula in Section 10.10.2.
   * AST and ALT ≤5 × institutional ULN at the time of randomization or pre-cytoreduction/general anesthesia;
   * Total bilirubin ≤1.5 × institutional ULN unless the participant has documented Gilbert's syndrome;
4. Prior history of thrombosis during corticosteroid use and/or asparaginase are eligible provided the patient receives anti-coagulant prophylaxis per institutional guidelines.
5. Cardiac shortening fraction ≥ 30% by echocardiogram or ejection fraction >50% by MUGA.

6 Participants with combined bone marrow and testicular relapse are eligible assuming orchiectomy is performed prior to randomization or is planned at the end of induction therapy.

5.2. Exclusion Criteria

1. Any history of prior or ongoing hepatic SOS or prior liver failure [defined as severe acute liver injury with encephalopathy and impaired synthetic function (INR of ≥1.5)].
2. Prior allo-HSCT or CAR T-cell therapy.
3. Isolated extramedullary leukemia.
4. Philadelphia-chromosome positive ALL, ie. BCR-ABL/t(9;22) present.
5. Prior therapy with a calicheamicin-conjugated antibody (eg, InO or gemtuzumab ozogamicin).
6. Participants with active, uncontrolled bacterial, fungal, or viral infection.
7. Hypersensitivity/allergy to both PEG-ASP and Erwinia-ASP

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2033-10-31 (Estimated); Study Completion 2036-11-04 (Estimated)

PRIMARY OUTCOMES:
Minimum Residual Disease (MRD) Negativity in participants achieving complete response (CR), complete response with incomplete platelet count recovery (CRp), or complete response with incomplete count recovery (CRi) | After 1 treatment cycle: Day 28 +/- 2 days
  MRD negativity status is determined based on the minimum MRD percentage between the date of CR/CRp/CRi and end of treatment test as assessed by RQ-PCR, with reflex to FC result if MRD is non-evaluable by RQ-PCR

SECONDARY OUTCOMES:
Event Free Survival (EFS) | From study start to first event (progression, relapse, failure to achieve CR/CRp/CRi by the end of induction, MRD persistence prior to HSCT [hematopoietic stem cell transplant], second malignancy, or death): up to 5 years from randomization
  EFS will be summarized using Kaplan-Meier methods and displayed graphically by treatment arm.
Duration of Response (DoR) for Participants Who Achieved CR/CRp/CRi | From date of first response to date of first event (objective progression, relapse as determined by investigator assessment, MRD persistence prior to HSCT, or death due to any cause, whichever occurs first): up to 5 years from End of Treatment
  DoR will be summarized using Kaplan-Meier methods.
Rate of hematopoietic stem cell transplantation (HSCT) | Up to 5 years from randomization
  HSCT rate will be summarized by descriptive analyses (ie, percentage of participants who underwent HSCT after treatment).
Overall Survival (OS) | From start of treatment to date of death due to any cause: up to 5 years from randomization
  OS will be summarized by treatment arm using Kaplan-Meier methods.
Number of participants reporting an Adverse Event (AE) | From time of informed consent up to a minimum of 60 calendar days after the last dose of study drug.
  The number and percentage of participants who experienced any AE, SAE (Serious Adverse Event), treatment related AE, and treatment related SAE will be summarized according to worst toxicity grades.
Pharmacokinetics (PK) parameter: InO Cmax | 1 treatment cycle: 28 days
  Descriptive summary statistics will be provided for InO serum concentrations at scheduled visits.
Number of Adverse Events (AE) reported by severity | From time of informed consent up to a minimum of 60 calendar days after the last dose of study drug.
  AEs will be graded by the investigator according to the CTCAE (Common Terminology Criteria for Adverse Events) version 4.03.
Pharmacokinetics (PK) parameter: InO trough levels | 1 treatment cycle: 28 days
  Descriptive summary statistics will be provided for InO serum concentrations at scheduled visits.
Rate of Chimeric antigen receptor (CAR) T-cell therapy | Up to 5 years from randomisation
  CAR T-cell therapy rate will be summarized by descriptive analyses (ie, the number, percent of participants who underwent CAR T-cell therapy after treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (74):
- St. Anna Kinderspital, Vienna, Austria
- Belgium (3):
  - Cliniques universitaires Saint-Luc, Brussels, Bruxelles-capitale, Région de
  - UZ Gent, Ghent, Oost-vlaanderen
  - UZ Leuven, Leuven, Vlaams-brabant
- Czechia (2):
  - Detska nemocnice FN Brno, Brno, Brno-město
  - Fakultni nemocnice v Motole, Prague
- Rigshospitalet, Copenhagen, Capital Region, Denmark
- Helsinki university hospital, Helsinki, Finland
- France (12):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice, Alpes-maritimes
  - CHU Strasbourg-Hautepierre, Service d'hematologie oncologie pediatrique, pediatrie 3, Strasbourg, Alsace
  - Bordeaux University Hospital - Pellegrin, Bordeaux, Aquitaine
  - CHU de Toulouse - Hôpital des Enfants - Hemato-Immuno-Oncologie, Toulouse, Haute-garonne
  - Hôpital Arnaud de Villeneuve - CHU Montpellier, Montpellier, Hérault
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Meurthe-et-moselle
  - Hôpital Jeanne de Flandre - CHRU, Lille, NORD
  - Assistance Publique - Hopitaux de Paris (AP-HP) - Hopital Robert Debre - Centre Hospitalo Universita, Paris, Paris
  - Institut d'Hématologie et d'Oncologie Pédiatrique, Lyon
  - CHU de Nantes - Hôpital Mère - Enfants, Nantes
  - Hôpital Armand Trousseau, Paris
  - CHRU De Rennes - Hôpital Sud, Rennes
- Germany (15):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Wuerzburg, Würzburg, Bavaria
  - Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
  - Charité Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitätsklinikum Gießen, Giessen
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
- Hungary (3):
  - Pécsi Tudományegyetem Klinikai Központ, Pécs, Baranya
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktatókórház, Miskolc, Borsod-Abauj Zemplen county
  - Semmelweis Egyetem, Budapest
- Israel (4):
  - Schneider Children's Medical Center, Petah Tikva, Central District
  - The Edmond and Lily Safra Children's Hospital; The Chaim Sheba Medical Center, Ramat Gan, Central District
  - Rambam Health Care Campus, Haifa, Northern District
  - Tel-Aviv Sourasky Medical Center Dana-Dwek Children's Hospital, Tel Aviv, TELL ABĪB
- Italy (11):
  - Azienda Ospedaliera di Rilievo Nazional Santobono Pausilipon, Napoli, Campania
  - IRCCS Istituto Giannina Gaslini, Genoa, Liguria
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardy
  - Ospedale Pediatrico Bambino Gesù IRCCS, Rome, ROMA
  - Policlinico "G. Rodolico", Catania, Sicily
  - Azienda Ospedale - Università Padova, Padua, Veneto
  - IRCCS - AOU di Bologna, Bologna
  - Azienda di Rilievo Nazionale e Alta Specializzazione Civico Di Cristina Benfratelli, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedale Regina Margherita, Torino
  - IRCCS Materno Infantile Burlo Garofolo, Trieste
- Prinses Maxima Centrum voor Kinderoncologie, Utrecht, Netherlands
- Norway (2):
  - Oslo Universitetssykehus Rikshospitalet, Oslo
  - Radium Hospital, Oslo
- Poland (2):
  - Szpital Uniwersytecki nr 1 im. dr. A. Jurasza w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw, Lower Silesian Voivodeship
- Narodny ustav detskych chorob, Bratislava, Bratislava Region, Slovakia
- Spain (9):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [LA Coruña]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona [barcelona]
  - Hospital Infantil Universitario Niño Jesús, Madrid, Madrid, Comunidad de
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Universitario La Paz, Madrid
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (3):
  - Skånes Universitetssjukhus Lund, Lund, Skåne LÄN [se-12]
  - Sahlgrenska Universitetssjukhuset Östra, Gothenburg, Västra Götalands LÄN [se-14]
  - Astrid Lindgrens Barnsjukhus, Stockholm
- Switzerland (3):
  - Inselspital Bern, Bern, Canton of Bern
  - CHUV (centre hospitalier universitaire vaudois), Lausanne, Canton of Vaud
  - Kinderspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1931036